CLINICAL TRIAL: NCT01262443
Title: Prospective Study to Evaluate the Acute and 6-month Efficacy of Transcatheter Radiofrequency Ablation of Common Atrial Flutter With a Standard Irrigated Catheter With Flexible Tip.
Brief Title: Efficacy of Transcatheter Radiofrequency Ablation of Atrial Flutter With Standard Irrigated Catheter With Flexible Tip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESREFO01
Record Dates: First submitted 2010-12-13; First posted 2010-12-17 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Flutter
Keywords: Atrial flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapy Cool Flex catheter group (Experimental): Therapy Cool Flex Catheter . No more available data
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Radiofrequency ablation by a standard 4mm irrigated flexible tip catheter

SUMMARY:
The purpose of this study is to evaluate the efficacy of transcatheter ablation of atrial flutter with a standard irrigated catheter with flexible tip, as evaluated by percentual success of the procedure.

DETAILED DESCRIPTION:
No more available data

ELIGIBILITY:
Inclusion Criteria:

* Both sexes; age>18 yrs
* ECG documentation of at least 2 episodes of common atrial flutter or evidence of ongoing atrial flutter.
* No contraindications to transcatheter radiofrequency ablation by a standard 4mm irrigated flexible tip catheter
* Patients willing to accept the tests and to follow standard procedures
* Patients who understand the nature of the procedure and who are willing to participate and to sign the informed consent before enrollment

Exclusion Criteria:

* Atrial fibrillation
* Any arrhythmia requiring antiarrhythmics in the 6 months post procedure
* Intra atrial thrombosis
* NYHA class IV
* Unstable Angina or Acute Myocardial Infarction (AMI) in the last 3 month
* Untreated Wolf Parkinson White syndrome
* Contraindications to oral anticoagulation
* Life expectancy < 12 month
* Major surgery or interventional procedure already planned in the 6 month following ablation
* Pregnancy or breast-feeding
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentual success of the procedure during the hospitalization | Up to 4 days
  Procedural success is defined as evidence of bidirectional block of cava tricuspidal istmus. The presence of block will be evaluated by mapping the electrical activation of the right atrium before and after pacing from thecoronary synus.
Percentual success of the procedure at 3 months from procedure | 3 months
  Procedural success is defined as evidence of bidirectional block of cava tricuspidal istmus. The presence of block will be evaluated by mapping the electrical activation of the right atrium before and after pacing from thecoronary synus.
Percentual success of the procedure at 6 months from procedure | 6 months
  Procedural success is defined as evidence of bidirectional block of cava tricuspidal istmus. The presence of block will be evaluated by mapping the electrical activation of the right atrium before and after pacing from thecoronary synus.

SECONDARY OUTCOMES:
•Synus rhythm maintenance in the absence of antiarrhythmics within 6 month from procedure. | Up to 4 days; 3-6 month
Duration of ablation procedure, number of radiofrequency erogations, duration and total energy given | Up to 4 days
Safety of the procedure | Up to 4 days
  recording of procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — Maria Cecilia Hospital
Locations (2):
- Italy (2):
  - Maria Cecilia Hospital, Cotignola, RA
  - Maria Pia Hospital, Torino, TO

IPD SHARING:
Plan to Share IPD: No